CLINICAL TRIAL: NCT06430112
Title: Liposomal Bupivacaine vs Ropivacaine for Ultrasound-guided Transversus Abdominis Plane Blocks in Laparoscopic Lower Abdominal Tumor Resection: A Prospective Randomized Trial
Brief Title: Liposomal Bupivacaine vs Ropivacaine for TAPBs
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ping Yu, Doctor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2023-485-01
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Abdominal Tumor; Postoperative Analgesia; Liposomal Bupivacaine; Ropivacaine
Keywords: liposomal bupivacaine; ropivacaine; transversus abdominis plane block; laparoscopic lower abdominal tumor resection; opioid consumption
MeSH Terms: conditions — Abdominal Neoplasms | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liposomal Bupivacaine group (Experimental): Liposomal Bupivacaine was used in the group
  Interventions: Drug: Liposomal Bupivacaine
- Ropivacaine group (Active Comparator): Ropivacaine was used in this group
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Liposomal Bupivacaine — After induction of anesthesia, bilateral TAPB was performed under ultrasound guidance. The patients in the bupivacaine liposome group were injected with bupivacaine liposome 133mg(10ml+ 10ml 0.9% normal saline mixed into 20ml)/ point (two points in total).
  Other Names: Bupivacaine liposome
  Arms: Liposomal Bupivacaine group
Drug: Ropivacaine — Patients in ropivacaine group were given 0.25% ropivacaine 20ml/ point (two points in total).
  Other Names: Ropivacaine Hydrochloride Injection
  Arms: Ropivacaine group

SUMMARY:
Few studies have compared the efficacy of ultrasound (US)-guided TAP blocks with Liposomal bupivacaine(LB) versus ropivacaine in reducing postoperative opioid usage in patients undergoing laparoscopic lower abdominal tumor Resection. Therefore, we are conducting this prospective, randomized controlled trial to compare the postoperative analgesic effects of LB and ropivacaine for TAP blocks among patients undergoing laparoscopic colorectal procedures.

DETAILED DESCRIPTION:
This study aimed to investigate the impact of liposomal bupivacaine (LB) on postoperative opioid usage for ultrasound(US)-guided transversus abdominis plane (TAP) blocks in laparoscopic colorectal resections. We divided 76 patients into two groups. An injection of bilateral TAP blocks was administered to LB group using 133mg liposomal bupivacaine in each block (266mg total), and to R group using 20 ml 0.25% ropivacaine in each block (40 ml total). Opioid consumption and pain scores at 6h, 24h, 48h and 72h were recorded postoperatively, as well as the total intraoperative remifentanil dose, the hospital stay lengths after surgery, and adverse events including dizziness, nausea, and vomiting.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing laparoscopic resection of lower abdominal tumors
2. ASA grade II-III
3. Age: 18-70 years.

Exclusion Criteria:

1. (1) The patient does not agree to participate in the clinical study
2. (2) The patient has a clear history of opioid tolerance or allergy
3. (3) The patient has a history of local anesthetic allergy
4. (4) Previous history of dementia, mental illness or other central nervous system diseases
5. (5) Have a history of chronic pain or are taking opioids and other analgesics
6. (6) Patients are generally in poor condition with a history of serious diseases of cardiovascular system, respiratory system, digestive system, urinary system or central nervous system, and may not survive for more than 3 months
7. (7) The patient had any of the following conditions in the 12 months before surgery: myocardial infarction, severe/unstable angina pectoris, coronary artery bypass grafting, congestive heart failure, cerebrovascular accident, pulmonary embolism
8. (8) Pregnant women
9. (9) Unable to cooperate with follow-up or poor compliance
10. (10) Patients with acute myocardial infarction, cardiac arrest or shock during surgery or hospitalization
11. (11) ASA score above grade III.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative opioid use | 3 days postoperatively
  The amount of drug used in the postoperative analgesia pump

SECONDARY OUTCOMES:
Postoperative pain score | 3 days postoperatively
  Postoperative VAS score
Postoperative adverse reactions | 3 days postoperatively
  Postoperative adverse reactions were followed up

CONTACTS AND LOCATIONS:
Overall Officials: Jingdun Xie, Principal Investigator — Department of Anesthesiology,Sun Yat-Sen University Cancer Center
Locations (1):
- Jingdun Xie, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
https://www.medicalresearch.org.cn/,Time: After completing the academic paper for publication
Supporting Information: Study Protocol
Time Frame: After completing the academic paper for publication
Access Criteria: The persons who were willing to study.